CLINICAL TRIAL: NCT04321135
Title: Avanzando Juntas: Adapting an Evidence Based Weight Loss Program for Hispanic Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Loyola University Chicago (Other)
Responsible Party: Principal Investigator, Melinda Stolley, Associate Director for Cancer Prevention and Control, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00030295
Record Dates: First submitted 2020-02-26; First posted 2020-03-25 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer; Gynecologic Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either a guided or self-guided lifestyle intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Lifestyle Program (Experimental): The Intervention will be conducted in a cohort of 20 (anticipated) and is designed to increase self-efficacy, social support and perceived access to healthy eating and exercise resources and promote weight loss. Participants assigned to the Guided Lifestyle Program will participate in twice weekly sessions - the first weekly session will be 120 minutes in length with the first hour addressing lifestyle change education and strategies. The second hour will be supervised exercise including aerobics and resistance training. The second weekly session will be a one-hour supervised exercise session. Participants will also receive 2-3 text messages weekly.They will also receive a participant informational binder with health and exercise information and tools as directed by ACS nutrition and physical activity guidelines.The Guided Lifestyle program is four months long (16 weeks). Please note, the Guided Lifestyle program participants will be offered a booster session off-study.
  Interventions: Behavioral: Guided Lifestyle Program Intervention
- Self-Guided Lifestyle Program (Active Comparator): In the self-guided weight loss program, participants will be given the sane informational binder with health and exercise information and tools as directed by ACS nutrition and physical activity guidelines but they will not receive in-person classes or text messaging. The study team will call these participants once a month to check in.
  Interventions: Behavioral: Self-Guided Lifestyle Program (Control Arm)

INTERVENTIONS:
Behavioral: Guided Lifestyle Program Intervention — The Guided Lifestyle Program will receive sessions that meet twice weekly and 2-3 text messages weekly.They will also receive a participant informational binder (wellness guide) with health and exercise information and tools as directed by ACS nutrition and physical activity guidelines.
  Arms: Guided Lifestyle Program
Behavioral: Self-Guided Lifestyle Program (Control Arm) — In the self-guided weight loss program, participants will be given the sane informational binder with health and exercise information and tools as directed by ACS nutrition and physical activity guidelines but they will not receive in-person classes or text messaging
  Arms: Self-Guided Lifestyle Program

SUMMARY:
This study examine the feasibility and efficacy of Avanzando Juntas, a four-month community-based lifestyle intervention rooted in the evidence-based Moving Forward lifestyle intervention developed with and for AA breast cancer survivors. This intervention was adapted in collaboration with Hispanic/Latina BC & GC survivors. It will offer twice-weekly sessions aimed at supporting adherence to ACS nutrition and physical activity guidelines to promote weight loss and improved quality of life.

DETAILED DESCRIPTION:
Aim 1. To adapt the Moving Forward weight loss intervention for overweight/obese Hispanic BCS using an iterative process engaging Hispanic BCS and a community advisory committee.

Aim 2. To conduct a randomized pilot with 40 overweight/obese Hispanic BCS to establish the feasibility of the adapted Moving Forward program based on recruitment, adherence, retention and efficacy.

Aim 3. To explore the effects of the adapted Moving Forward program (Avanzando Juntas) on anthropometric (weight, % body fat, lean mass), behavioral (dietary intake, physical activity) psychosocial (quality of life) and biological (cholesterol, hemoglobin A1c, adiponectin, leptin, inflammation, insulin resistance) outcomes.

Hypothesis: Women in the weight loss program will exhibit improvements in outcomes compared to women in the wait list control group.

Avanzando Juntas supports BC & GC survivors in adopting physical activity and eating patterns to promote weight loss, bolster QOL and reduce the risk for comorbidities and, potentially, BC & GC recurrence. A strong, multidisciplinary study team provides expertise in culturally competent programs for Hispanic BCS, cognitive behavioral lifestyle interventions, body composition, breast cancer and program adaptation.

This study is novel in its focus on weight loss among Hispanic BCS and the incorporation of anthropometric, behavioral, biological and psychosocial outcomes. An additional strength is the foundation of community partnerships that will support the current study's efforts, as well as those for a larger trial, and, if successful, the dissemination of the program.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identify as Hispanic or Latina
2. Female
3. Stage 0 -III Breast and Gynecological cancer survivors
4. Treatment (surgery, chemotherapy and/or radiation) completed at least three months before recruitment (ongoing hormonal therapy is acceptable)
5. Age >18 at time of diagnosis
6. BMI at least 25 kg/m2 BMI between 25 and 55 - chosen because this will include only those participants who are overweight and would not be harmed by a 5% weight loss

Exclusion Criteria:

1. Plans to move from the community during the study
2. A medical condition limiting adherence to diet or physical activity components
3. History of significant mental illness
4. Currently pregnant, less than 3 months post-partum, or pregnancy anticipated during the study
5. Taking any medications prescribed by a doctor to lose weight participate in any organized weight loss programs or has undergone weight loss surgery or planning to undergo weight loss surgery in the next year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female Breast and Gynecological study participants
Enrollment: 40 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Change in body composition | Baseline to 4 month
  Ratio of percent lean mass to percent adiposity as measured by Bio-electrical Impedance Analysis Scale. More lean mass and less adiposity is favorable
Change in intake of fruits and vegetables | Baseline to 4 month
  ASA24 dietary analysis of self reported food consumption
Change of intake of red meat/processed meat | Baseline to 4 month
  ASA24 dietary analysis of self reported food consumption
Change in levels of physical activity- minutes per week | Baseline to 4 month
  Change of ActiGraph monitored activity
Change in levels of physical activity- #times per week | Baseline to 4 month
  Change of ActiGraph monitored activity
Change in resistance training- Handgrip strength | Baseline to 4 month
  Jamar Plus Digital Hand Dynamometer
Change in resistance training- Strength and endurance | Baseline to 4 month
  30-Second Chair Stand (Sit to Stand)
Change in Quality of Life- PROMIS (Patient Reported Outcomes Measurement Information System) | Baseline to 4 month
  Patient Reported Outcomes Measurement Information System (PROMIS) T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. PROMIS measures physical function, depression, anxiety, fatigue, sleep disturbance, social roles, pain interference, social isolation, cognitive function, support, self-efficacy and sexual function. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like pain interference, a T-score of 60 is one SD worse than average. By comparison, a pain interference T-score of 40 is one SD better than average.
Changes in Systolic and Diastolic Blood Pressure | Baseline to 4 month
  Participants systolic and diastolic blood pressure will be measured using a digital, automated unit
Change in Biomarkers- Lipids | Baseline to 4 month
  Lipid blood tests measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers- Glycohem | Baseline to 4 month
  Glycohem blood tests measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers- Glucose | Baseline to 4 month
  Glucose blood tests measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers- C-Peptide | Baseline to 4 month
  C-Peptide blood tests measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers- Insulin | Baseline to 4 month
  Insulin blood tests measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers- hs CRP | Baseline to 4 month
  hs CRP blood tests measured by Wisconsin Diagnostic Laboratory
Change in Biomarkers-Adipokines- Adiponectin | Baseline to 4 month
  Adiponectin blood tests
Change in Biomarkers-Adipokines- Leptin | Baseline to 4 month
  Adiponectin blood tests
Change in waist circumference | Baseline to 4 month
  Change in waist circumference measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States